CLINICAL TRIAL: NCT04074330
Title: Phase 1/2 Study of TAK-981 in Combination With Rituximab in Patients With Relapsed/Refractory CD20-Positive Non-Hodgkin Lymphoma
Brief Title: A Study of TAK-981 Given With Rituximab in Adults With Relapsed or Refractory CD20-Positive Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrolment Challenges
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-981-1501; U1111-1236-0243 (Registry Identifier: WHO); 2020-003946-36 (EudraCT Number)
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — TAK-981; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Phase 1: TAK-981 10mg QW (Experimental): Participants with indolent or aggressive non-Hodgkin lymphoma (NHL) received TAK-981 10 mg, infusion, intravenously (IV), once weekly (QW) on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 milligram per square meter (mg/m^2), infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or disease progression (PD) or unacceptable toxicity.
  Interventions: Drug: TAK-981; Drug: Rituximab
- Phase 1: TAK-981 40mg QW (Experimental): Participants with indolent or aggressive NHL received TAK-981 40 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
  Interventions: Drug: TAK-981; Drug: Rituximab
- Phase 1: TAK-981 60mg QW (Experimental): Participants with indolent or aggressive NHL received TAK-981 60 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
  Interventions: Drug: TAK-981; Drug: Rituximab
- Phase 1: TAK-981 90mg QW (Experimental): Participants with indolent or aggressive NHL received TAK-981 90 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
  Interventions: Drug: TAK-981; Drug: Rituximab
- Phase 1: TAK-981 90mg BIW (Experimental): Participants with indolent or aggressive NHL received TAK-981 90 mg, infusion, IV, BIW on Days 1, 4, 8, and 11 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
  Interventions: Drug: TAK-981; Drug: Rituximab
- Phase 1: TAK-981 120mg QW (Experimental): Participants with indolent or aggressive NHL received TAK-981 120 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
  Interventions: Drug: TAK-981; Drug: Rituximab
- Phase 1: Japan Lead-in: TAK-981 60mg QW (Experimental): Japanese participants with indolent or aggressive NHL received TAK-981 60 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
  Interventions: Drug: TAK-981; Drug: Rituximab
- Phase 1: Japan Lead-in: TAK-981 60mg BIW (Experimental): Japanese participants with indolent or aggressive NHL received TAK-981 60 mg, infusion, IV, BIW on Days 1, 4, 8, and 11 every 21 days in each 21-day treatment cycle for up to 12 months or PD or unacceptable toxicity.
  Interventions: Drug: TAK-981
- Phase 2 (A): TAK-981 120 mg (Experimental): Participants with relapsed or refractory (r/r) diffuse large B-cell lymphoma (DLBCL) received TAK-981 120 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab infusion, intravenously, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
  Interventions: Drug: TAK-981; Drug: Rituximab
- Phase 2 (C): TAK-981 120 mg (Experimental): Participants with follicular lymphoma (FL) received TAK-981 120 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab infusion, intravenously, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
  Interventions: Drug: TAK-981; Drug: Rituximab

INTERVENTIONS:
Drug: TAK-981 — TAK-981 intravenous infusion.
Drug: Rituximab — Rituximab intravenous infusion.
  Arms: Phase 1: Japan Lead-in: TAK-981 60mg QW; Phase 1: TAK-981 10mg QW; Phase 1: TAK-981 120mg QW; Phase 1: TAK-981 40mg QW; Phase 1: TAK-981 60mg QW; Phase 1: TAK-981 90mg BIW; Phase 1: TAK-981 90mg QW; Phase 2 (A): TAK-981 120 mg; Phase 2 (C): TAK-981 120 mg

SUMMARY:
This study is about a medicine called TAK-981 given with rituximab, used to treat adults with relapsed or refractory CD20-positive non-Hodgkin lymphoma.

This study has 2 parts.

The main aims of the study are:

* To check for side effects from treatment with TAK-981 given with rituximab.
* To check how much TAK-981 participants can tolerate.
* To check if participants with diffuse large B-cell lymphoma or follicular lymphoma respond well to treatment.

Participants will receive TAK-981 and rituximab in 21-day cycles. They will continue treatment for about 12 months unless their condition gets worse (disease progression), they cannot tolerate the treatment, or they leave the study for certain reasons.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-981 in combination with rituximab. The study will include a dose escalation phase (Phase 1) and an expansion phase in select non-Hodgkin lymphoma (NHL) indications (Phase 2).

The study will enroll approximately 180 participants, approximately 35 participants in Phase 1 and approximately 145 participants in Phase 2. The participants with indolent or aggressive relapsed or refractory (r/r) NHL in Phase 1 will identify the maximum tolerated dose (MTD) and/or pharmacologically active dose (PAD). PAD can be defined retrospectively once MTD is reached and it can below MTD or coincide with it. In the dose escalation phase, the starting dose of TAK-981 will be 10 mg. The RP2D will be determined based on the available safety, preliminary pharmacokinetic (PK), pharmacodynamic information data, and after any early antitumor activity observed along with the statistical inference from the Bayesian logistic regression modeling (BLRM).

Participants in the Phase 2 will be enrolled once the Phase 1 of the study is completed, and MTD and/or PAD is determined. Phase 2 will explore the efficacy and safety of TAK-981 in combination with rituximab in participants with select NHL types and indications. Participants in Phase 2 will be enrolled in one of the three treatment arms based on Cohorts:

* Phase 2, Cohort A r/r DLBCL Progressed after CAR T-cell therapy:TAK-981+Rituximab
* Phase 2, Cohort B:r/r DLBCL;no CAR T-cell Therapy;2-3 Prior Lines: Two Dose Levels of TAK-981+Rituximab
* Phase 2, Cohort C:r/r FL;no CAR T-cell Therapy;2-3 Prior Lines: Two Dose Levels of TAK-981+Rituximab

This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 72 months. Participants will make multiple visits to the clinic, and will attend the end of treatment (EOT) visit 30 days after receiving their last dose of drug or before the start of subsequent systemic anticancer therapy, whichever occurs first for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all the following inclusion criteria to be enrolled in the study:

1. Participant Population:

   o. For Phase 1 Dose Escalation: o. aNHL including mantle cell lymphoma and DLBCL histologies such as transformed DLBCL from low-grade lymphoma (follicular or others), DLBCL associated with small-cell infiltration in bone marrow, B-cell lymphoma with intermediate features between DLBCL and Burkitt's lymphoma or with intermediate features between DLBCL and Hodgkin lymphoma, FL grade 3B, and aggressive B-cell lymphoma unclassifiable who must have previously received rituximab, cyclophosphamide, doxorubicin (hydroxydaunorubicin), vincristine, (Oncovin) and prednisone (R-CHOP) (or equivalent anti-CD20 containing therapy) and 1 additional line of therapy in the r/r setting.

   o. iNHL (including FL of grades 1-3A and marginal zone lymphoma) refractory to rituximab or to any other anti-CD20 monoclonal antibodies, who have received at least 1 prior systemic therapy for r/r iNHL.

   o. Rituximab or anti-CD20 refractoriness is defined as failure to respond to, or progression during, any previous rituximab/anti-CD20-containing regimen (monotherapy or combined with chemotherapy), or progression within 6 months of the last rituximab or anti-CD20 dose.

   Note: The minimum qualifying rituximab/anti-CD20 dose is 1 full cycle (that is, weekly*4 doses monotherapy or 1 complete dose if combined with chemotherapy). Prior anti-CD20 antibody or cytotoxic drugs may have been administered as single agents or as components of combination therapies. Each repeated course of the same single-agent or combination is considered an independent regimen.

   o. For Phase 2, the following confirmed CD20+: o. r/r DLBCL progressed or relapsed after a prior CAR T-cells therapy that has received approval by a health authority for the treatment of DLBCL (Cohort A).

   o. r/r DLBCL that has progressed or relapsed after at least 2 but no more than 3 prior lines of systemic therapy and has not I prior cellular therapy. At least one prior line of therapy must have included a CD20-targeted therapy (Cohort B).

   o. r/r FL that has progressed or relapsed after at least 2 but no more than 3 prior lines of systemic therapy. At least 1 prior line of therapy must have included a CD20-targeted therapy (Cohort C).
2. Must be considered ineligible in the opinion of the investigator, or refused autologous stem-cell transplantation (ASCT).
3. Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to (<=) 2.
4. Adequate bone marrow function per local laboratory reference range at screening as follows:

   o Platelet count greater than or equal to (>=) 75.0*10^9/L, Grade 2 thrombocytopenia (platelet count >=50.0*10^9 per liter [/L]) is allowed if it is clearly due to marrow involvement with no evidence of myelodysplastic syndrome or hypoplastic bone marrow if found. Absolute neutrophil count (ANC) >=1.0*10^9/L. Hemoglobin >=85 gram per liter (g/L) (red blood cell [RBC] transfusion allowed >=14 days before assessment).
5. Adequate renal and hepatic function, per local laboratory reference range at screening as follows:

   * Calculated creatinine clearance >=30 milliliter per minute (mL/min) calculated with Cockcroft-Gault formula.
   * Potassium levels >=lower limit of normal (LLN). For potassium >upper limit of normal (ULN) discussion with Takeda medical monitor (MM)/designee recommended.
   * Aspartate aminotransferase and alanine aminotransferase <=3.0*the ULN of the institution's normal range; bilirubin <=1.5*ULN. Participants with Gilbert's syndrome may have a bilirubin level >1.5*ULN, per discussion between the investigator and the medical monitor.
6. Left ventricular ejection fraction (LVEF) >=40 percent (%); as measured by echocardiogram or multiple gated acquisition (MUGA) scan.
7. Suitable venous access for safe drug administration and the study-required PK and pharmacodynamic sampling.
8. Have at least 1 bidimensionally measurable lesion per Lugano Classification by computed tomography (CT). Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
9. Willing to consent to 1 mandatory pretreatment and 1 on-treatment skin biopsy during Phase 1. The skin biopsy entry requirement may be discontinued by the sponsor once there is enough pharmacodynamic evidence of target engagement.
10. For participants enrolled in Phase 2, if available, mandatory submission of archival tumor tissue acquired ≤12 months prior to screening.
11. Recovered to Grade 1, baseline or established as sequela, from all toxic effects of previous therapy (except alopecia, neuropathy, autoimmune endocrinopathies with stable endocrine replacement therapy, neurotoxicity [Grade 1 or 2 permitted], or bone marrow parameters [any of Grade 1, 2, permitted if directly related to bone marrow involvement]).

Exclusion Criteria:

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Central nervous system lymphoma; active brain or leptomeningeal metastases, as indicated by positive cytology from lumbar puncture or CT scan/magnetic resonance imaging (MRI).
2. History of Grade >=3 infusion-related reaction (IRR) that lead to permanent discontinuation of previous rituximab treatment.
3. Post transplantation lymphoproliferative disease except relapsed NHL after ASCT.
4. Undergone ASCT or treatment with cellular therapy including CAR T within <=12 weeks of TAK-981 dosing.
5. Prior allogeneic hematopoietic stem-cell transplantation.
6. Lymphomas with leukemic expression.
7. Prior anticancer therapy including chemotherapy, hormonal therapy, or investigational agents within 2 weeks or within at least 5 half-lives before TAK-981 dosing, whichever is shorter. Low dose steroids (oral prednisone or equivalent <=20 mg per day), hormonal therapy for prostate cancer or breast cancer (in adjuvant situation), and treatment with bisphosphonates and receptor activator of nuclear factor kappa-B ligand (RANKL) inhibitors are allowed.
8. Major surgery within 14 days before the first dose of study drug and not recovered fully from any complications from surgery.
9. Significant medical diseases or conditions, as assessed by the Investigators and sponsor that would substantially increase the risk-benefit ratio of participating in the study. This includes but is not limited to acute myocardial infarction or unstable angina within the last 6 months; uncontrolled diabetes mellitus; significant active bacterial, viral, or fungal infections; severely immunocompromised state; severe non-compensated hypertension and congestive heart failure New York Heart Association Class III or IV; ongoing symptomatic cardiac arrhythmias of >Grade 2, pulmonary embolism, or symptomatic cerebrovascular events; or any other serious cardiac condition (example, pericardial effusion or restrictive cardiomyopathy). Chronic atrial fibrillation on stable anticoagulant therapy is allowed.
10. Known chronic hepatitis C and/or positive serology (unless due to vaccination or passive immunization due to immunoglobulin [Ig] therapy) for chronic hepatitis B. Known Human Immunodeficiency Virus (HIV) infection.
11. Second malignancy within the previous 3 years, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, cervical carcinoma in situ, resected colorectal adenomatous polyps, breast cancer in situ, or other malignancy for which the participant is not on active anticancer therapy.
12. Receipt of any live vaccine within 4 weeks of initiation of study treatment.
13. Active, uncontrolled autoimmune disease requiring >20 mg of prednisone or equivalent, cytotoxics or biologicals.
14. Corticosteroid use within 1 week before the first dose of study drug, except as indicated for other medical conditions such as inhaled steroid for asthma, topical steroid use, or as premedication for administration of study drug or contrast. Participants requiring steroids at daily doses >20 mg prednisone equivalent systemic exposure daily, or those who are administered steroids for lymphoma control or white blood cell count lowering are not eligible.
15. With baseline prolongation of the QT interval with Fridericia correction method (QTcF) (example, >470 milliseconds (ms) for women and >450 ms for men and a history of congenital long QT syndrome, or torsades de pointes).
16. Receiving or requiring the continued use of medications that are known to be strong or moderate inhibitors and inducers of Cytochrome P450 3A4/5 (CYP3A4/5) and strong P-glycoprotein (Pgp) inhibitors. To participate in this study, such participants should discontinue use of such agents for at least 2 weeks (1 week for CYP3A4/5 and Pgp inhibitors) before receiving a dose of TAK-981.
17. Participants in Germany who are committed to an institution by virtue of an order issued either by judicial or administrative authorities as per German law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (59):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic - Cancer Center - Rochester - PPDS, Rochester, Minnesota
  - Levine Cancer Institute - Charlotte, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - City of Hope - Comprehensive Cancer Center (CCC), Portland, Oregon
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Texas Oncology (Medical City) - USOR, Dallas, Texas
  - Texas Oncology (Tyler) - USOR, Tyler, Texas
- Canada (2):
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Sir Mortimer B Davis Jewish General Hospital, Pointe-Claire, Quebec
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
- France (8):
  - Institut Paoli Calmettes, Marseille, Bouches-du-Rhone
  - Hopital Francois Mitterand, Dijon, Cote-d'Or
  - CHU Montpellier - Hopital St Eloi, Montpellier, Herault
  - Hopital Prive Sevigne, Rennes, Ille-et-Vilaine
  - Hotel Dieu - Nantes, Nantes, Loire-Atlantique
  - Centre Henri Becquerel, Rouen, Seine-Maritime
  - Hopital Saint Antoine, Paris
  - Hopital Universitaire Pitie Salpetriere, Paris
- Germany (8):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitatsklinikum Tubingen, Tübingen, Baden-Wurttemberg
  - Klinikum rechts der Isa der Technischen Universitaet Muenchen, München, Bavaria
  - Universitatsklinikum Wurzburg, Würzburg, Bavaria
  - Universitatsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Otto-von-Guericke-Universitat Magdeburg, Magdeburg, Saxony-Anhalt
  - Charite - Universitatsmedizin Berlin, Berlin
- Italy (9):
  - Azienda Ospedaliera Cardinale G Panico, Tricase, Apulia
  - Azienda Sanitaria Locale di Ravenna, Ravenna, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Istituto Nazionale Dei Tumori, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda, Milan, Lombardy
  - A.O.U. Maggiore della Carita, Novara, Piedmont
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Turin, Piedmont
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
- Japan (5):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aiti
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National University Corporation Tohoku University Tohoku University Hospital, Sendai, Miyagi
  - Kindai University Hospital, Osakasayama-Shi, Osaka
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Koto-Ku, Tokyo
- Spain (7):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Complejo Asistencial Universitario de Salamanca H. Clinico, Salamanca
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- United Kingdom (6):
  - Derriford Hospital, Plymouth, Devon
  - Beatson West of Scotland Cancer Centre - PPDS, Glasgow, Lanarkshire
  - University College London, London, London, City of
  - Royal Marsden Hospital - Downs Road, London, London, City of
  - Oxford University Hospitals NHS Trust, Oxford, Oxfordshire
  - University Hospital Birmingham, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Nakamura A, Grossman S, Song K, Xega K, Zhang Y, Cvet D, Berger A, Shapiro G, Huszar D. The SUMOylation inhibitor subasumstat potentiates rituximab activity by IFN1-dependent macrophage and NK cell stimulation. Blood. 2022 May 5;139(18):2770-2781. doi: 10.1182/blood.2021014267. PMID 35226739
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a352

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in the United States, Canada, and Japan from 15 October 2019 to 26 April 2023.
Pre-assignment Details: Participants with a diagnosis of Non-Hodgkin Lymphoma were enrolled in this study consisting of Phase 1 (Dose Escalation and Japan-Specific lead-in cohorts), and Phase 2 (Dose Expansion) to receive TAK-981 and/or rituximab.
Groups:
- Japan Lead-in: TAK-981 60mg QW: Japanese participants with indolent or aggressive NHL received TAK-981 60 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Japan Lead-in: TAK-981 60mg BIW: Japanese participants with indolent or aggressive NHL received TAK-981 60 mg, infusion, IV, BIW on Days 1, 4, 8, and 11 every 21 days in each 21-day treatment cycle for up to 12 months or PD or unacceptable toxicity.
Period: Dose Escalation (up to 19.36 Months)
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg
Started | 3 | 4 | 3 | 7 | 8 | 6 | 1 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 3 | 7 | 8 | 6 | 1 | 3 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 0 | 0 | 5 | 2 | 2 | 1 | 2 | 0 | 0
Not completed — Start of New Systemic Treatment | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Period: Dose Expansion (up to 42 Months)
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set consisted of participants who have received at least 1 dose, even if incomplete, of study drug.
Groups:
- Phase 1: TAK-981 10mg QW: Participants with indolent or aggressive NHL received TAK-981 10 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Japan Lead-in: TAK-981 60mg BIW: Participants with indolent or aggressive NHL received TAK-981 60 mg, infusion, IV, BIW on Days 1, 4, 8, and 11 every 21 days in each 21-day treatment cycle for up to 12 months or PD or unacceptable toxicity.
- Phase 2 (A): TAK-981 120 mg: Participants with r/r DLBCL received TAK-981 120 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab infusion, intravenously, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Phase 2 (C): TAK-981 120 mg: Participants with FL received TAK-981 120 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab infusion, intravenously, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg | Total
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 8 | 6 | 1 | 3 | 2 | 1 | 38
Age, Continuous [Mean (Full Range); unit: years] | 64.0 [56.0 to 77.0] | 69.3 [60.0 to 80.0] | 73.0 [67.0 to 79.0] | 57.7 [29.0 to 65.0] | 64.8 [46.0 to 78.0] | 58.8 [35.0 to 79.0] | 61.0 [61.0 to 61.0] | 70.3 [68.0 to 72.0] | 71 [67 to 75] | 55 [55 to 55] | 64.5 [29.0 to 80.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 3 | 0 | 0 | 12
  Male | 2 | 3 | 2 | 5 | 6 | 5 | 0 | 0 | 2 | 1 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 2 | 7 | 7 | 6 | 1 | 3 | 2 | 1 | 36
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 3 | 3 | 3 | 7 | 6 | 6 | 0 | 0 | 2 | 1 | 31
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With One or More Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse event (AE) means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product. A TEAE was defined as an adverse event which occurred on or after the first dose of study drug and no more than 30 days after the last dose of study drug.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 42 months)
Population: Safety Analysis Set consisted of participants who have received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 8 | 6 | 1 | 3
Participants | 3 | 4 | 3 | 6 | 8 | 6 | 1 | 3

2. Primary Outcome: Phase 1: Number of Participants With Grade 3 or Higher TEAEs
Description: AE means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product whether or not it is related to the medicinal product. A TEAE was defined as an adverse event which occurred on or after the first dose of study drug and no more than 30 days after the last dose of study drug. A severity grade was evaluated as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0, except for Cytokine Release Syndrome (CRS), which was assessed by American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading criteria.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 42 months)
Population: Safety Analysis Set consisted of participants who have received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 8 | 6 | 1 | 3
Participants | 1 | 4 | 1 | 2 | 7 | 3 | 1 | 2

3. Primary Outcome: Phase 1: Duration of TEAEs
Description: AE means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product whether or not it is related to the medicinal product. A TEAE was defined as an adverse event which occurred on or after the first dose of study drug and no more than 30 days after the last dose of study drug. As per planned analysis, data for this outcome measure were collected and analyzed for the combined population (Phase 1: TAK-981 60mg QW+Japan Lead-in: TAK-981 60mg QW) based on regimen in which same dose groups in Phase 1 irrespective of nationality were pooled.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 42 months)
Population: Safety Analysis Set consisted of participants who have received at least 1 dose, even if incomplete, of study drug.
Measure: Median (Full Range); unit: days
Groups:
- Phase 1 + Japan Lead-in: TAK-981 60mg QW: Participants with indolent or aggressive NHL received TAK-981 60 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity. All participants who received TAK-981 60 mg QW in Phase 1 irrespective of nationality were pooled.
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1 + Japan Lead-in: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 4 | 7 | 8 | 6 | 3
days | 57.0 [1 to 775] | 8.0 [1 to 575] | 13.0 [1 to 473] | 2.0 [1 to 360] | 11.0 [1 to 274] | 10.0 [1 to 838] | 2.0 [1 to 657]

4. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs) Per Dose Level
Description: DLTs were evaluated according to NCI CTCAE, Version 5.0.
Time Frame: Up to 42 months
Population: The DLT-evaluable analysis set will include participants enrolled in the Phase 1 portion of the study who experienced a DLT at any time after initiation of the first infusion of TAK-981 or who completed all planned infusions of TAK-981 as per schedule plus 3 infusions of rituximab without experiencing a DLT. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 4 | 6 | 1 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved complete response (CR) and partial response (PR), as defined by the investigator according to Lugano classification for lymphomas during the study.
Time Frame: Up to 42 months
Population: Response-evaluable analysis set consisted of participants who have received at least 1 dose of study drug, have sites of measurable disease at Baseline, and 1 postbaseline disease assessment, or were discontinued due to symptomatic deterioration or death before a postbaseline evaluation happens.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg
Number analyzed (Participants) | 2 | 1
percentage of participants | 50 | 100

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-981
Description: As per planned analysis, data for this outcome measure were collected and analyzed for the combined population (Phase 1: TAK-981 60mg QW+Japan Lead-in: TAK-981 60mg QW) based on regimen in which same dose groups in Phase 1 irrespective of nationality were pooled. This outcome measure was planned to be analyzed for Phase 1 only.
Time Frame: Cycle 1: Days 1 and 8, pre-infusion and at multiple timepoints (Up to 24 hours) post end of infusion (cycle length=21 days)
Population: Pharmacokinetic (PK) analysis set consisted of participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Overall number of participants analyzed is the number of participants available for analysis. Number of participants analyzed is the number of participants available for analysis during the specified time-point.
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/ml)
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1 + Japan Lead-in: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 4 | 7 | 7 | 6 | 3
nanograms per millilitre (ng/ml)
  Cycle 1 Day 1 | 39.8 (19.1) | 184 (139) | 444 (323) | 648 (214) | 810 (305) | 740 (491) | 833 (73.3)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4 | 6 | 5 | 6 | 3
  Cycle 1 Day 8 | 51.4 (13.9) | 200 (152) | 595 (410) | 600 (146) | 967 (299) | 981 (272) | 731 (346)

7. Secondary Outcome: Tmax: Time of First Occurrence of the Maximum Plasma Concentration (Cmax) for TAK-981
Description: as for outcome 6
Time Frame: as for outcome 6
Population: PK analysis set consisted of participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Overall number of participants analyzed is the number of participants available for analysis. Number of participants analyzed is the number of participants available for analysis during the specified time-point.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1 + Japan Lead-in: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 4 | 7 | 7 | 6 | 3
hours
  Cycle 1 Day 1 | 1.17 [1.15 to 1.20] | 1.15 [1.14 to 1.42] | 1.14 [0.97 to 1.29] | 1.14 [1.09 to 1.39] | 1.17 [1.07 to 1.53] | 1.28 [1.10 to 1.95] | 1.12 [1.12 to 1.48]
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4 | 6 | 5 | 6 | 3
  Cycle 1 Day 8 | 1.15 [1.07 to 1.24] | 1.08 [1.04 to 1.27] | 0.95 [0.93 to 1.02] | 1.08 [1.02 to 1.72] | 1.05 [1.00 to 1.30] | 1.11 [1.05 to 1.19] | 1.12 [1.04 to 1.67]

8. Secondary Outcome: AUC0-t: Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for TAK-981
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1 + Japan Lead-in: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 4 | 7 | 7 | 6 | 3
hours*ng/mL
  Cycle 1 Day 1 | 146 (15.0) | 477 (130) | 1070 (456) | 1310 (380) | 1490 (475) | 1640 (484) | 1520 (103)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4 | 6 | 5 | 6 | 3
  Cycle 1 Day 8 | 140 (25.6) | 517 (236) | 1160 (510) | 1290 (351) | 1640 (483) | 1780 (333) | 1420 (356)

9. Secondary Outcome: AUC0-∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-981
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h.ng/ml
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1 + Japan Lead-in: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 4 | 7 | 6 | 6 | 3
h.ng/ml
  Cycle 1 Day 1 | 151 (15.1) | 498 (128) | 1110 (465) | 1360 (398) | 1640 (445) | 1600 (550) | 1560 (114)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4 | 6 | 5 | 6 | 3
  Cycle 1 Day 8 | 150 (19.2) | 538 (242) | 1210 (514) | 1330 (359) | 1780 (490) | 1830 (344) | 1460 (382)

10. Secondary Outcome: t1/2z: Terminal Disposition Phase Half-life for TAK-981
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1 + Japan Lead-in: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 4 | 7 | 6 | 6 | 3
hours
  Cycle 1 Day 1 | 5.06 [4.78 to 5.41] | 5.88 [5.31 to 6.76] | 6.02 [5.67 to 6.46] | 5.75 [4.50 to 7.01] | 4.88 [4.21 to 7.23] | 5.78 [2.87 to 8.35] | 5.91 [5.12 to 6.00]
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4 | 6 | 5 | 6 | 3
  Cycle 1 Day 8 | 5.03 [3.15 to 5.92] | 5.92 [5.51 to 6.15] | 5.77 [5.12 to 7.14] | 5.78 [4.98 to 6.29] | 5.59 [3.10 to 10.93] | 5.73 [5.23 to 6.46] | 5.45 [4.16 to 6.91]

11. Secondary Outcome: CL: Total Clearance After Intravenous Administration for TAK-981
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: litres per hour (L/h)
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1 + Japan Lead-in: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 4 | 7 | 6 | 6 | 3
litres per hour (L/h)
  Cycle 1 Day 1 | 66.8 (6.37) | 83.8 (17.8) | 65.2 (37.0) | 72.7 (27.2) | 58.2 (15.5) | 81.8 (24.7) | 38.6 (2.78)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4 | 6 | 5 | 6 | 3
  Cycle 1 Day 8 | 67.4 (8.23) | 75.2 (43.8) | 57.8 (26.2) | 73.3 (25.9) | 53.9 (14.6) | 68.0 (16.1) | 43.2 (13.1)

12. Secondary Outcome: Vss: Volume of Distribution at Steady State After Intravenous Administration for TAK-981
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: litres (L)
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1 + Japan Lead-in: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 4 | 7 | 6 | 6 | 3
litres (L)
  Cycle 1 Day 1 | 396 (72.8) | 517 (202) | 406 (277) | 352 (136) | 255 (75.5) | 410 (156) | 154 (1.72)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4 | 6 | 5 | 6 | 3
  Cycle 1 Day 8 | 352 (79.9) | 456 (278) | 332 (211) | 347 (110) | 273 (201) | 307 (95.0) | 189 (68.0)

13. Secondary Outcome: Phase 1: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved CR and PR, as defined by the investigator according to Lugano classification for lymphomas during the study.
Time Frame: Up to 42 months
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 6 | 6 | 1 | 3
percentage of participants | 33.3 | 50.0 | 66.7 | 14.3 | 0 | 33.3 | 0 | 33.3

14. Secondary Outcome: Phase 1: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants who achieved CR, PR, and stable disease (SD) as defined by the investigator according to Lugano classification for Lymphomas during the study.
Time Frame: Up to 42 months
Population: as for outcome 5
Measure: Number; unit: percenage of participants
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 6 | 6 | 1 | 3
percenage of participants | 100 | 50.0 | 100 | 28.6 | 16.7 | 50.0 | 0 | 33.3

15. Secondary Outcome: Phase 1: Duration of Response (DOR)
Description: DOR is the time from the date of first documentation of a PR or better to the date of first documentation of PD for responders (PR or better). DOR was assessed by the investigator according to Lugano classification for lymphoma during the study.
Time Frame: Up to 42 months
Population: Response-evaluable analysis set consisted of participants who have received at least 1 dose of study drug, have sites of measurable disease at Baseline, and 1 postbaseline disease assessment, or were discontinued due to symptomatic deterioration or death before a postbaseline evaluation happens. Overall number of participants analyzed is the number of participants with events.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
months | 8.31 [8.31 to 8.31] |  |  | 2.73 [2.73 to 2.73] |  |  |  | 8.94 [8.94 to 8.94]

16. Secondary Outcome: Phase 1: Time to Progression (TTP)
Description: TTP is defined as the time from the date of first study drug administration to the date of first documented disease progression. TTP was assessed by the investigator according to Lugano classification for lymphoma during the study.
Time Frame: Up to 42 months
Population: as for outcome 15
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 2 | 0 | 0 | 5 | 4 | 2 | 0 | 1
months | 12.42 [2.69 to 12.42] |  |  | 1.58 [0.95 to 3.98] | 1.48 [0.00 to 3.91] | NA [0.92 to 19.09] — Median was not estimable as there were censored participants with events. |  | 13.18 [13.18 to 13.18]

17. Secondary Outcome: Phase 1: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of the first dose administration to the date of first documentation of PD or death due to any cause, whichever occurs first. PD was determined by Response Evaluation Criteria in Lymphoma. PFS was assessed by the investigator according to Lugano classification for lymphoma during the study.
Time Frame: Up to 42 months
Population: Response-evaluable analysis set consisted of participants who have received at least 1 dose of study drug, have sites of measurable disease at Baseline, and 1 postbaseline disease assessment, or were discontinued due to symptomatic deterioration or death before a postbaseline evaluation happens. Overall number of participants analyzed are the number of participants with events.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 2 | 0 | 0 | 5 | 4 | 2 | 0 | 1
months | 12.42 [2.69 to 12.42] |  |  | 1.58 [1.25 to 3.98] | 2.33 [0.43 to 3.91] | NA [1.61 to 19.09] — Median was not estimable as there were censored participants with events. |  | 13.18 [13.18 to 13.18]

18. Secondary Outcome: Phase 1: Fold Change From Baseline in Levels of TAK-981-Small Ubiquitin-like Modifier (TAK-981-SUMO) Adduct Formation in Blood as Assessed by Flow Cytometry During Phase 1
Description: The level of TAK-981-SUMO adduct formation was evaluated as the percentage of adduct formed in blood. Positive change denotes improvement.
Time Frame: Cycle 1 Day 1 (1 hour, 4 hours, 8 hours) and Day 8 (Pre-dose, 1 hour, 4 hours and 8 hours) (Cycle length = 21 days)
Population: Pharmacodynamic analysis set consisted of participants who have provided evaluable blood samples (C1D1 predose sample and at least 1 postdose sample). Number of participants available is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 5 | 5 | 1 | 3
ratio
  Cycle 1 Day 1 /1 Hour Postdose | 4.1 (0.54) | 5.7 (1.47) | 6.3 (1.02) | 9.5 (1.04) | 7.6 (0.73) | 9.9 (2.84) | 4.9 (NA) — Standard deviation was not estimable as there was only one participant. | 6.7 (1.42)
  Cycle 1 Day 1 /4 Hours Postdose: number analyzed (Participants) | 3 | 4 | 3 | 7 | 5 | 2 | 0 | 1
  Cycle 1 Day 1 /4 Hours Postdose | 3.6 (0.66) | 4.7 (1.18) | 4.7 (1.28) | 6.7 (1.07) | 4.9 (1.69) | 6.5 (0.56) |  | 4.1 (NA) — Standard deviation was not estimable as there was only one participant.
  Cycle 1 Day 1 /8 Hours Postdose: number analyzed (Participants) | 3 | 4 | 3 | 7 | 5 | 4 | 1 | 3
  Cycle 1 Day 1 /8 Hours Postdose | 3.7 (0.27) | 4.5 (1.22) | 4.1 (1.24) | 5.6 (1.05) | 4.6 (0.72) | 5.2 (0.64) | 3.0 (NA) — Standard deviation was not estimable as there was only one participant. | 3.3 (0.32)
  Cycle 1 Day 8 /Predose: number analyzed (Participants) | 3 | 4 | 3 | 6 | 4 | 5 | 1 | 3
  Cycle 1 Day 8 /Predose | 1.8 (0.13) | 1.9 (0.68) | 1.9 (0.27) | 2.5 (0.88) | 2.8 (0.51) | 2.8 (1.50) | 1.1 (NA) — Standard deviation was not estimable as there was only one participant. | 1.6 (0.17)
  Cycle 1 Day 8 /1 Hour Postdose: number analyzed (Participants) | 3 | 4 | 3 | 5 | 4 | 5 | 1 | 3
  Cycle 1 Day 8 /1 Hour Postdose | 4.6 (0.19) | 6.6 (0.96) | 8.0 (0.87) | 9.1 (3.21) | 7.8 (0.61) | 11.6 (6.34) | 5.0 (NA) — Standard deviation was not estimable as there was only one participant. | 5.4 (0.69)
  Cycle 1 Day 8 /4 Hours Postdose: number analyzed (Participants) | 3 | 4 | 3 | 6 | 4 | 2 | 0 | 1
  Cycle 1 Day 8 /4 Hours Postdose | 3.9 (0.19) | 6.2 (1.87) | 5.1 (0.70) | 6.1 (2.16) | 5.8 (0.65) | 5.6 (1.73) |  | 4.3 (NA) — Standard deviation was not estimable as there was only one participant.
  Cycle 1 Day 8 /8 Hours Postdose: number analyzed (Participants) | 3 | 4 | 3 | 6 | 4 | 5 | 1 | 3
  Cycle 1 Day 8 /8 Hours Postdose | 3.2 (0.55) | 4.2 (1.34) | 4.0 (0.49) | 5.3 (1.97) | 4.0 (1.43) | 7.1 (2.83) | 2.9 (NA) — Standard deviation was not estimable as there was only one participant. | 3.3 (0.38)

19. Secondary Outcome: Phase 1: Levels of TAK-981-Small Ubiquitin-like Modifier (TAK-981-SUMO) Adduct Formation in Skin as Assessed by Immunohistochemistry (IHC) During Phase 1
Description: The level of TAK-981-SUMO adduct formation was evaluated as the percentage of adduct formed in skin.
Time Frame: Cycle 1 Days 1 and 8 (Cycle length = 21 days)
Population: Pharmacodynamic analysis set consisted of participants who have provided evaluable skin biopsies (screening sample and postdose sample). Overall number of participants available is the number of participants available for analysis. Number of participants available is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: % adduct positive
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 1 | 4 | 1 | 3
% adduct positive
  Cycle 1 Day 1 /Predose: number analyzed (Participants) | 3 | 4 | 3 | 6 | 0 | 4 | 1 | 3
  Cycle 1 Day 1 /Predose | 0.0 (0.03) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) |  | 0.0 (0.0) | 0.0 (NA) — Standard deviation was not estimable as there was only one participant. | 0.0 (0.0)
  Cycle 1 Day 8 | 1.2 (1.15) | 15.8 (12.70) | 27.0 (12.29) | 22.6 (9.47) | 59.7 (NA) — Standard deviation was not estimable as there was only one participant. | 11.2 (11.35) | 1.4 (NA) — Standard deviation was not estimable as there was only one participant. | 29.5 (19.88)

20. Secondary Outcome: Phase 1: Fold Change From Baseline in SUMO Pathway Inhibition in Blood as Assessed by Flow Cytometry During Phase 1
Description: SUMO pathway inhibition in blood was evaluated by flow cytometry with an antibody recognizing SUMO2/3 chains.
Time Frame: Cycle 1 Day 1 (1 hour, 4 hours, 8 hours) and Day 8 (Pre-dose, 1 hour, 4 hours and 8 hours) (Cycle length = 21 days)
Population: Pharmacodynamic analysis set consisted of participants who have provided evaluable blood samples (C1D1 predose sample and at least 1 postdose sample). Overall number of participants analyzed are the number of participants available for analysis. Number of participants available is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 5 | 5 | 1 | 3
ratio
  Cycle 1 Day 1 /1 Hour Postdose | 0.9 (0.05) | 0.8 (0.15) | 0.5 (0.36) | 0.6 (0.11) | 0.5 (0.26) | 0.6 (0.22) | 0.1 (NA) — Standard deviation was not estimable as there was only one participant. | 0.8 (0.33)
  Cycle 1 Day 1 /4 Hours Postdose: number analyzed (Participants) | 3 | 4 | 3 | 7 | 5 | 2 | 0 | 1
  Cycle 1 Day 1 /4 Hours Postdose | 0.9 (0.07) | 0.8 (0.15) | 0.5 (0.34) | 0.5 (0.15) | 0.4 (0.30) | 0.9 (0.14) |  | 1.0 (NA) — Standard deviation was not estimable as there was only one participant.
  Cycle 1 Day 1 /8 Hours Postdose: number analyzed (Participants) | 3 | 4 | 3 | 7 | 5 | 4 | 1 | 3
  Cycle 1 Day 1 /8 Hours Postdose | 1.0 (0.05) | 0.8 (0.17) | 0.5 (0.33) | 0.5 (0.15) | 0.5 (0.22) | 0.7 (0.28) | 0.2 (NA) — Standard deviation was not estimable as there was only one participant. | 0.8 (0.24)
  Cycle 1 Day 8 /Predose: number analyzed (Participants) | 3 | 4 | 3 | 6 | 4 | 5 | 1 | 3
  Cycle 1 Day 8 /Predose | 0.9 (0.09) | 1.1 (0.37) | 0.8 (0.12) | 1.1 (0.46) | 0.9 (0.07) | 1.1 (0.25) | 0.2 (NA) — Standard deviation was not estimable as there was only one participant. | 0.7 (0.33)
  Cycle 1 Day 8 /1 Hour Postdose: number analyzed (Participants) | 3 | 4 | 3 | 5 | 4 | 5 | 1 | 3
  Cycle 1 Day 8 /1 Hour Postdose | 0.9 (0.10) | 0.8 (0.34) | 0.5 (0.19) | 0.5 (0.05) | 0.5 (0.14) | 0.6 (0.10) | 0.1 (NA) — Standard deviation was not estimable as there was only one participant. | 0.5 (0.25)
  Cycle 1 Day 8 /4 Hours Postdose: number analyzed (Participants) | 3 | 4 | 3 | 6 | 4 | 2 | 0 | 1
  Cycle 1 Day 8 /4 Hours Postdose | 0.9 (0.09) | 0.7 (0.31) | 0.5 (0.23) | 0.6 (0.20) | 0.7 (0.05) | 0.7 (0.10) |  | 1.2 (NA) — Standard deviation was not estimable as there was only one participant.
  Cycle 1 Day 8 /8 Hours Postdose: number analyzed (Participants) | 3 | 4 | 3 | 6 | 4 | 5 | 1 | 3
  Cycle 1 Day 8 /8 Hours Postdose | 0.9 (0.09) | 0.7 (0.37) | 0.5 (0.04) | 0.5 (0.13) | 0.5 (0.35) | 0.7 (0.17) | 0.2 (NA) — Standard deviation was not estimable as there was only one participant. | 0.7 (0.31)

21. Secondary Outcome: Phase 1: SUMO Pathway Inhibition in Skin as Assessed by Immunohistochemistry (IHC) During Phase 1
Description: SUMO pathway inhibition in skin was evaluated with skin tissue biopsies by IHC.
Time Frame: Cycle 1 Days 1 and 8 (Cycle length = 21 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: % Sumo 2/3 positive
Arm/Group | Phase 1: TAK-981 10mg QW | Phase 1: TAK-981 40mg QW | Phase 1: TAK-981 60mg QW | Phase 1: TAK-981 90mg QW | Phase 1: TAK-981 90mg BIW | Phase 1: TAK-981 120mg QW | Japan Lead-in: TAK-981 60mg QW | Japan Lead-in: TAK-981 60mg BIW
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 1 | 4 | 1 | 3
% Sumo 2/3 positive
  Cycle 1 Day 1 /Predose: number analyzed (Participants) | 3 | 4 | 3 | 6 | 0 | 4 | 1 | 3
  Cycle 1 Day 1 /Predose | 83.40383 (2.692876) | 87.74383 (5.142812) | 89.60727 (5.528530) | 89.63755 (4.044536) |  | 75.79235 (2.586486) | 86.85370 (NA) — Standard deviation was not estimable as there was only one participant. | 69.65077 (19.035919)
  Cycle 1 Day 8 | 82.26130 (2.017705) | 79.34405 (10.262143) | 55.69903 (19.325964) | 52.54200 (15.606775) | 51.84200 (NA) — Standard deviation was not estimable as there was only one participant. | 63.14625 (15.415286) | 69.68880 (NA) — Standard deviation was not estimable as there was only one participant. | 41.79763 (21.796849)

22. Secondary Outcome: Phase 2: Number of Participants With One or More Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 1
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 42 months)
Population: Safety Analysis Set consisted of participants who have received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

23. Secondary Outcome: Phase 2: Number of Participants With Grade 3 or Higher TEAEs
Description: as for outcome 2
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 42 months)
Population: Safety Analysis Set consisted of participants who have received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

24. Secondary Outcome: Phase 2: Duration of TEAEs
Description: AE means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product whether or not it is related to the medicinal product. A TEAE was defined as an adverse event which occurred on or after the first dose of study drug and no more than 30 days after the last dose of study drug.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 42 months)
Population: Safety Analysis Set consisted of participants who have received at least 1 dose, even if incomplete, of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg
Number analyzed (Participants) | 2 | 1
days | 8.0 [1 to 483] | 2.0 [1 to 349]

25. Secondary Outcome: Phase 2: Disease Control Rate (DCR)
Description: CR is defined as the percentage of participants who achieved CR, PR, and SD as defined by the investigator according to Lugano classification for Lymphomas during the study.
Time Frame: Up to 42 months
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg
Number analyzed (Participants) | 2 | 1
percentage of participants | 1 | 1

26. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: as for outcome 15
Time Frame: Up to 42 months
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg
Number analyzed (Participants) | 2 | 1
months | 3.32 [3.32 to 3.32] | 0.03 [0.03 to 0.03]

27. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: as for outcome 16
Time Frame: Up to 42 months
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg
Number analyzed (Participants) | 2 | 1
months | 5.32 [5.32 to 5.32] | 1.48 [1.48 to 1.48]

28. Secondary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: as for outcome 17
Time Frame: Up to 42 months
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2 (A): TAK-981 120 mg | Phase 2 (C): TAK-981 120 mg
Number analyzed (Participants) | 2 | 1
months | 3.15 [1.0 to 5.3] | 1.48 [1.48 to 1.48]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 42 months)
Description: Safety Analysis Set consisted of participants who have received at least 1 dose, even if incomplete, of study drug.
Groups:
- Phase 1: TAK981 10mg QW: Participants with indolent or aggressive NHL received TAK-981 10 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Phase 1: TAK981 40mg QW: Participants with indolent or aggressive NHL received TAK-981 40 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Phase 1: TAK981 60mg QW: Participants with indolent or aggressive NHL received TAK-981 60 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Phase 1: TAK981 90mg QW: Participants with indolent or aggressive NHL received TAK-981 90 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Phase 1: TAK981 90mg BIW: Participants with indolent or aggressive NHL received TAK-981 90 mg, infusion, IV, BIW on Days 1, 4, 8, and 11 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Phase 1: TAK981 120mg QW: Participants with indolent or aggressive NHL TAK-981 120 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Japan Lead-in: TAK981 60mg QW: Japanese participants with indolent or aggressive NHL received TAK-981 60 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab 375 mg/m^2, infusion, IV, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Japan Lead-in: TAK981 60mg BIW: Japanese participants with indolent or aggressive NHL received TAK-981 60 mg, infusion, IV, BIW on Days 1, 4, 8, and 11 every 21 days in each 21-day treatment cycle for up to 12 months or PD or unacceptable toxicity.
- Phase 2 (A): TAK981 120mg: Participants with r/r DLBCL received TAK-981 120 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab infusion, intravenously, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
- Phase 2 (C): TAK981 120mg: Participants with FL received TAK-981 120 mg, infusion, IV, QW on Days 1 and 8 every 21 days in each 21-day treatment cycle in combination with rituximab infusion, intravenously, once on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of each 21-day treatment cycle from Cycle 2 for up to 12 months or PD or unacceptable toxicity.
Arm/Group | Phase 1: TAK981 10mg QW | Phase 1: TAK981 40mg QW | Phase 1: TAK981 60mg QW | Phase 1: TAK981 90mg QW | Phase 1: TAK981 90mg BIW | Phase 1: TAK981 120mg QW | Japan Lead-in: TAK981 60mg QW | Japan Lead-in: TAK981 60mg BIW | Phase 2 (A): TAK981 120mg | Phase 2 (C): TAK981 120mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/4 | 0/3 | 1/7 | 4/8 | 1/6 | 0/1 | 0/3 | 1/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/4 | 1/3 | 2/7 | 5/8 | 2/6 | 0/1 | 0/3 | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 6/7 | 8/8 | 6/6 | 1/1 | 3/3 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: TAK981 10mg QW (N=3) | Phase 1: TAK981 40mg QW (N=4) | Phase 1: TAK981 60mg QW (N=3) | Phase 1: TAK981 90mg QW (N=7) | Phase 1: TAK981 90mg BIW (N=8) | Phase 1: TAK981 120mg QW (N=6) | Japan Lead-in: TAK981 60mg QW (N=1) | Japan Lead-in: TAK981 60mg BIW (N=3) | Phase 2 (A): TAK981 120mg (N=2) | Phase 2 (C): TAK981 120mg (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: TAK981 10mg QW (N=3) | Phase 1: TAK981 40mg QW (N=4) | Phase 1: TAK981 60mg QW (N=3) | Phase 1: TAK981 90mg QW (N=7) | Phase 1: TAK981 90mg BIW (N=8) | Phase 1: TAK981 120mg QW (N=6) | Japan Lead-in: TAK981 60mg QW (N=1) | Japan Lead-in: TAK981 60mg BIW (N=3) | Phase 2 (A): TAK981 120mg (N=2) | Phase 2 (C): TAK981 120mg (N=1)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Campylobacter colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 3 | 3 | 5 | 0 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 2 | 2 | 0 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram P wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 1 | 2 | 5 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 4 | 1 | 0 | 3 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Infusion site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 4 | 0 | 1 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 5 | 3 | 5 | 1 | 2 | 2 | 1
QRS axis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Testicular oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to enrollment challenges.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT04074330/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT04074330/SAP_001.pdf